CLINICAL TRIAL: NCT07248150
Title: Perceptions of Healthcare Professionals Toward Clinical Pharmacy Practice in Egypt: A Cross-Sectional Observational Survey (Sub-Study of the Ph.D. Protocol "Role of Clinical Pharmacy and Mobile Medical Applications in Detection and Minimization of Medication Errors in Hospitalized Patients From Adults and Children")
Brief Title: Perceptions of Healthcare Professionals Toward Clinical Pharmacy Practice in Egypt
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Mohammed Abd Elhamid Mohammed Tony, clinical pharmacist and PHD researcher, Beni-Suef University
Other Study IDs: FMBSUREC/03102023/Tony
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Perception of Clinical Pharmacy Practice
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare Professionals Survey Group
  Interventions: Other: Survey Questionnaire

INTERVENTIONS:
Other: Survey Questionnaire — A structured, self-administered questionnaire developed by the research team to assess healthcare professionals' perceptions, attitudes, and level of trust toward clinical pharmacy practice in hospital settings. The survey was distributed both online and in paper form across different hospitals in Egypt. No clinical or therapeutic intervention was performed.

SUMMARY:
This study aims to explore how healthcare professionals in Egypt perceive the role of clinical pharmacists within hospital practice. It is an observational cross-sectional survey designed to gather opinions and attitudes toward clinical pharmacy services. The information collected will help identify areas that can improve collaboration between pharmacists and other healthcare team members and support future development of clinical pharmacy practice in Egypt.

ELIGIBILITY:
Inclusion Criteria:

Healthcare professionals currently working in hospital settings in Egypt.

Includes physicians, pharmacists, nurses, and physical therapists.

Participants aged 18 years or older.

Willing to voluntarily complete the study questionnaire (online or paper form).

Exclusion Criteria:

Individuals not belonging to the healthcare team.

Students, administrative staff, or non-clinical workers.

Participants younger than 18 years old.

Incomplete or duplicate survey responses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study included healthcare professionals working in Egyptian hospitals, such as physicians, pharmacists, nurses, and physical therapists. All participants were adults aged 18 years or older and voluntarily completed a structured questionnaire designed to assess their perceptions and attitudes toward clinical pharmacy practice.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Perception Score Toward Clinical Pharmacy Practice | from July 2024 to October 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy - Beni-Suef University, Cairo (Beni Suef Site), Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset includes responses from healthcare professionals collected under confidentiality agreements. Only summarized and anonymized results will be published in scientific journals.